CLINICAL TRIAL: NCT02554968
Title: Reliability and Validity of Five Shoulder-Specific Patient Reported Outcome Measures for Use in Patients With Head and Neck Cancer
Brief Title: Reliability and Validity of Patient Reported Outcome Measures in Head and Neck Cancer
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Melissa M. Eden, PT, DPT, OCS, Mayo Clinic
Other Study IDs: 15-005266
Record Dates: First submitted 2015-09-16; First posted 2015-09-18 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Shoulder Pain; Head and Neck Cancer
MeSH Terms: conditions — Shoulder Pain; Head and Neck Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study participants: Study participants will complete study related documents including a demographics questionnaire and the shoulder-related patient reported outcome measures.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires

SUMMARY:
This study will utilize Rasch analysis to study the construct validity and reliability of five shoulder-related patient-reported outcome measures in patients reporting shoulder impairment following surgery for head and neck cancer.

DETAILED DESCRIPTION:
This study is a cross-sectional, questionnaire-based psychometric study. The purpose of the study is to: (1) use Rasch methodology to assess the reliability, construct validity, and overall appropriateness of test score interpretation of 5 shoulder-related patient reported outcome measures in patients experiencing shoulder dysfunction following neck dissection surgery for head and neck cancer; and (2) based on these findings, provide recommendations of which patient reported outcome measure or combination of measures most accurately reflects shoulder disability in patients who experience shoulder dysfunction following neck dissection surgery. Two-hundred and fifty subjects will be recruited during regularly scheduled clinical visits at Mayo Clinic. Subjects will complete five shoulder-related patient reported outcome measures on only one occasion, therefore subjects will be responsible for study participation only at the time of enrollment and same day completion of study-related documents. Upon the conclusion of data collection, Rasch analysis will be utilized to analyze data related to the research objectives, and descriptive statistics will be utilized to describe the sample.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral or bilateral neck dissection procedure for management of head and neck cancer within the past 2 weeks to 18 months
* Endorse some level of shoulder impairment (Answer "yes" when asked "are you currently experiencing any shoulder weakness or discomfort as a result of your surgery?")
* 18-90 years of age
* Adequate fluency in the English language to complete the study-related forms and questionnaires

Exclusion Criteria:

• No reported shoulder impairment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients reporting shoulder discomfort, stiffness or weakness following a neck dissection procedure for management of head and neck cancer.
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2015-09; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Disability of the Arm, Shoulder and Hand | One day
QuickDASH | One day
Shoulder Pain and Disability Index | One day
University of Washington Quality of Life Scale (shoulder-subscale) | One day
Neck Dissection Impairment Index | One day

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Mayo Clinic, Phoenix, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- [Derived] Eden MM, Kunze KL, Galantino ML, Kolber MJ, Cheng MS. Shoulder-Specific Patient-Reported Outcome Measures for Use in Patients With Head and Neck Cancer: An Assessment of Reliability, Construct Validity, and Overall Appropriateness of Test Score Interpretation Using Rasch Analysis. Phys Ther. 2021 Nov 1;101(11):pzab160. doi: 10.1093/ptj/pzab160. PMID 34174083